CLINICAL TRIAL: NCT00930033
Title: Randomized Phase III Trial Evaluating the Importance of Nephrectomy in Patients Presenting With Metastatic Renal Cell Carcinoma Treated With Sunitinib
Brief Title: Clinical Trial to Assess the Importance of Nephrectomy
Acronym: CARMENA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pfizer (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P070144
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Nephrectomy,; metastatic renal cell carcinoma,; sunitinib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nephrectomy; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Nephrectomy + sunitinib
  Interventions: Procedure: Nephrectomy
- B (Experimental): Sunitinib alone
  Interventions: Other: Sunitinib alone

INTERVENTIONS:
Procedure: Nephrectomy — Current surgery
  Arms: A
Other: Sunitinib alone — Sunitinib alone without nephrectomy
  Other Names: Sunitinib alone without nephrectomy
  Arms: B

SUMMARY:
The study compare the standard treatment with nephrectomy + sunitinib to treatment with sunitinib alone without nephrectomy. This study will be the first trial on this competitive context

DETAILED DESCRIPTION:
The 2 previous studies on the impact of nephrectomy (EORTC, SWOG) in metastatic renal cell carcinoma have justified recommendation to initial nephrectomy for patients presenting with metastatic renal cell carcinoma. But these studies were performed at the time of immunotherapy.

The objective is Evaluation of the importance of nephrectomy in patients with metastatic renal cell carcinoma treated with sunitinib (AA) Arm A : Nephrectomy followed by Sunitinib Arm B : Sunitinib alone Sunitinib will be administrated orally daily for 4 weeks followed by a 2 week rest( schedule 4/2), 6 weeks are considered as a cycle The starting dose will be 50 mg daily with provision for dose reduction based on tolerability Patient will be treated until disease progression or unacceptable toxicity occurrence or withdraw.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* ECOG Performance Status 0 - 1
* Biopsy (primary tumour or metastases) confirming the diagnosis of clear cell carcinoma
* Documented metastatic disease
* Absence of prior systemic treatment for kidney cancer including AA
* Tumour amenable to nephrectomy (partial or total) in the opinion of the patient's urologist. Patients presenting with an inferior vena cava thrombosis can be included.
* Patients for which the indication of Sunitinib is considered according to the recommendations rules given by national health authorities of participating countries. The prescription of Sunitinib in the circumstances of the study is considered as a standard treatment.
* Platelets > or = 100 x 109/L, haemoglobin >or = 9 g/dl, neutrophils >or = 1.5 x 109/L;
* Bilirubin < or = 2 mg/dL, aspartate transaminase (ASAT) and alanine transaminase (ALAT)< or = 2.5 times the upper normal limit (UNL) or < or = 5 times UNL for patients with liver metastases
* Patients of child bearing age should use contraceptive methods
* Patient able to follow the procedures outlined in the protocol as far as the planning of visits and examinations are concerned.
* Life expectancy ≥ 3 months
* Written informed consent
* Patient without brain metastases or with radiotherapy or surgery treated brain metastases without progression into 6 weeks and non treated by corticoid
* Patient non treated by anticoagulants excepted HBPM

Exclusion Criteria:

* Prior systemic treatment for kidney cancer (including Anti Angiogenic)
* Bilateral kidney cancer
* Pregnant or breast feeding women
* Acute coronary syndrome or episode of myocardial infarction or severe or unstable angina within the last 6 months as well as severe diabetes with severe peripheral arteriopathy or deep phlebitis not treated with low molecular weight heparin or arterial thrombosis within the last 3 months
* Patients being treated with antivitamin K with curative intent (please note that patients being treated with low molecular weight heparin can be included)
* Medical, general or psychiatric difficulties which, in the opinion of the Investigator, would make it inappropriate for trial entry
* Symptomatic or untreated brain metastases (patients with brain metastases that have been treated by radiotherapy or surgery and have stable disease within 6 weeks, and are not requiring treatment with corticosteroids can be included)
* Previous history of gastric disease or malabsorption, syndrome compromising the absorption of Sunitinib
* Experimental treatment within the 28 days preceding inclusion
* Other cancer within the previous 5 years (except for insitu skin carcinoma and treated localised prostate cancer with undetectable PSA)
* Patient has received treatment with IV biphosphonate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2009-09-09 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is overall survival. | starting at 4 months

SECONDARY OUTCOMES:
Objective Response (complete or partial) is evaluated according to RECIST 1.1 criteria | Starting at 4 months
Clinical benefit (complete response, partial or stable for at least 12 weeks). | Starting at 4 months
Progression-Free Survival | Starting at 4 months
Non-compliance to Sunitinib treatment is evaluated in arm A (nephrectomy + sunitinib) as the percentage of patients not starting sunitinib treatment within 6 weeks after nephrectomy | Starting at 4 months
Non-compliance to sunitinib treatment is evaluated in arm B (sunitinib alone) as the percentage of patients needing nephrectomy | Starting at 4 months
Post operative morbidity is evaluated as the percentage of deaths within 30 days following nephrectomy | Starting at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Mejean, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Necker, Paris, France

REFERENCES:
- [Background] Mejean A, Ravaud A, Thezenas S, Chevreau C, Bensalah K, Geoffrois L, Thiery-Vuillemin A, Cormier L, Lang H, Guy L, Gravis G, Rolland F, Linassier C, Lechevallier E, Oudard S, Laguerre B, Gross-Goupil M, Bernhard JC, Colas S, Albiges L, Lebret T, Treluyer JM, Timsit MO, Escudier B. Sunitinib Alone or After Nephrectomy for Patients with Metastatic Renal Cell Carcinoma: Is There Still a Role for Cytoreductive Nephrectomy? Eur Urol. 2021 Oct;80(4):417-424. doi: 10.1016/j.eururo.2021.06.009. Epub 2021 Jun 27. PMID 34187771
- [Background] Mejean A, Ravaud A, Thezenas S, Colas S, Beauval JB, Bensalah K, Geoffrois L, Thiery-Vuillemin A, Cormier L, Lang H, Guy L, Gravis G, Rolland F, Linassier C, Lechevallier E, Beisland C, Aitchison M, Oudard S, Patard JJ, Theodore C, Chevreau C, Laguerre B, Hubert J, Gross-Goupil M, Bernhard JC, Albiges L, Timsit MO, Lebret T, Escudier B. Sunitinib Alone or after Nephrectomy in Metastatic Renal-Cell Carcinoma. N Engl J Med. 2018 Aug 2;379(5):417-427. doi: 10.1056/NEJMoa1803675. Epub 2018 Jun 3. PMID 29860937
- [Derived] Leon L, Garcia-Figueiras R, Suarez C, Arjonilla A, Puente J, Vargas B, Mendez Vidal MJ, Sebastia C. Recommendations for the clinical and radiological evaluation of response to treatment in metastatic renal cell cancer. Target Oncol. 2014 Mar;9(1):9-24. doi: 10.1007/s11523-013-0304-7. Epub 2013 Dec 12. PMID 24338498